CLINICAL TRIAL: NCT04722016
Title: LUNG ULTRASONOGRAPHY DECREASES RADIATION EXPOSURE
Acronym: LUDRE
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, associate professor, Hacettepe University
Other Study IDs: GO-LUNG
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Newborn Rds; Transient Tachypnea of the Newborn; Pneumonia
Keywords: lung ultrasonography; chest x ray; newborn
MeSH Terms: conditions — Pulmonary Atelectasis; Transient Tachypnea of the Newborn; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aimed to decrease in the number of chest X-rays in newborns with respiratory distress, with the use of lung ultrasonography.

From January 2019 to June 2020, 104 newborn infants with respiratory distress enrolled in this study. We used bed side ultrasound as the first line tecnique for lung imaging. X-ray were taken in cases with increasing respiratory distress in spite of treatment according to diagnosis depending on USG findings. We calculated decreased number of chest X-ray for every patient and evaluated the estimated decrease in radiation exposure.

DETAILED DESCRIPTION:
Background:

Chest X-ray is commonly used as first line imaging method to diagnose the reason of respiratory distress in NICUs. Lung ultrasound is a new diagnostic tool for lung imaging, and this method has been used more common recently in NICUs.

Objectives:

We aimed to determine the decrease in the number of chest X-rays in newborns with respiratory distress, with the use of lung ultrasonography.

Methods:

From January 2019 to June 2020, 104 newborn infants with respiratory distress enrolled in this study. We used bed side ultrasound as the first line tecnique for lung imaging. X-ray were taken in cases with increasing respiratory distress in spite of treatment according to diagnosis depending on USG findings. We calculated decreased number of chest X-ray for every patient and evaluated the estimated decrease in radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Term or preterm neonates with respiratory distress that started within the first 24 h after birth were included if they showed at admission signs of respiratory distress defined as: tachypnea (respiratory rate >60 breaths/min), intercostal/subcostal retractions, grunting, or FiO2 requirement >0.21.

Exclusion Criteria:

* Patients with a diagnosis of major malformations or chromosomal abnormalities, inherited metabolic diseases, congenital muscle disease-hypotonicity, hypoxic ischemic encephalopathy were not enrolled.

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term or preterm neonates with respiratory distress that started within the first 24 h after birth
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Reduced radiation exposure | 18 months
  We aimed to decrease in the number of chest X-rays in newborns with respiratory distress, with the use of lung ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escourrou G, De Luca D. Lung ultrasound decreased radiation exposure in preterm infants in a neonatal intensive care unit. Acta Paediatr. 2016 May;105(5):e237-9. doi: 10.1111/apa.13369. No abstract available. PMID 26880491
- [Derived] Tandircioglu UA, Yigit S, Oguz B, Kayki G, Celik HT, Yurdakok M. Lung ultrasonography decreases radiation exposure in newborns with respiratory distress: a retrospective cohort study. Eur J Pediatr. 2022 Mar;181(3):1029-1035. doi: 10.1007/s00431-021-04296-5. Epub 2021 Oct 23. PMID 34687334
- See also: lung ultrasonography — https://pubmed.ncbi.nlm.nih.gov/30957609/